CLINICAL TRIAL: NCT01941849
Title: A Phase I Trial of Vandetanib Combined With 131I-mIBG Radiotherapy in Patients With Neuroendocrine Tumours, Advanced Phaeochromocytoma and Paraganglioma
Brief Title: Phase I Trial of Vandetanib Combined With 131I-mIBG to Treat Patients With Advanced Phaeochromocytoma and Paraganglioma
Acronym: VIBRaNT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor patient accrual
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0499
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Phaeochromocytoma; Paraganglioma
Keywords: Phaeochromocytoma; Paraganglioma; Neuroendocrine Tumour; Vandetanib; 131I-mIBG; Radionucleotide Therapy; Vascular Endothelial Growth Factor (VEGF); Epidermal Growth Factor Receptor (EGFR); RET; Tyrosine Kinase
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neuroendocrine Tumors | interventions — vandetanib; 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib + 131I-mIBG (Experimental): Vandetanib (100, 200 or 300 mg once daily) in combination with 131I-mIBG radiation therapy (activity to be prescribed to deliver whole body absorbed dose of 0.5 Gy) on day 1 of each 12-weekly cycle.
  Patients will receive up to 4 cycles of vandetanib in combination with 131I-mIBG.
  Interventions: Drug: Vandetanib; Radiation: 131I-mIBG

INTERVENTIONS:
Drug: Vandetanib — 100 mg, 200 mg or 300 mg taken once a day during each 12-weekly cycle
  Other Names: Caprelsa
Radiation: 131I-mIBG — Activity will be prescribed to deliver whole body absorbed dose of 0.5 Gy (+/-10%)
  Other Names: Iodine-131 labelled Meta-iodobenzylguanine

SUMMARY:
The phase I trial aims to determine the recommended phase II dose (RP2D) of vandetanib in combination with standard radiation therapy, 131I-mIBG, in patients with advanced phaeochromocytoma (phaeo) and paraganglioma (PG) by assessing the safety and tolerability of the combination treatment.

DETAILED DESCRIPTION:
VIBRaNT is a registered phase I trial in patients with locally advanced or metastatic phaeochromocytoma or paraganglioma, not amenable to surgical resection.

Patients will receive vandetanib (an inhibitor of VEGF, EGFR and RET tyrosine kinase) in combination with standard radiation therapy Iodine-131 labelled Meta-iodobenzylguanidine (131I-mIBG).

Vandetanib and 131I-mIBG will be given in 12-weekly cycles: 131I-miBG will be given on day 1 of each cycle and vandetanib will started on day 1 of each cycle and continue to be taken once every day. The phase I trial aims to determine with recommended phase II dose of vandetanib (either 100, 200 or 300 mg once daily) - the dose of vandetanib that patients will receive will depend on the dose under investigation at the time of patient registration.

The vandetanib dose will be determined by the Modified Continual Reassessment Method (mCRM) - a toxicity model which described the probability of a toxicity occurring at each dose level, which is based on clinical judgement and any available toxicity data.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological/cytological diagnosis of advanced phaeo/PG defined as patients with local or metastatic disease not amenable to surgical resection, or R1 resection post original surgical debulking
2. Positive 123I-mIBG diagnostic scan
3. Stable blood pressure (<140/90mmHg), if appropriate, on anti-hypertensive therapy
4. No previous systemic chemotherapy within 3 months prior to registration
5. No previous mIBG therapy within 12 months prior to registration (previous cumulative activity must not exceed 15 GBq)
6. Measurable disease (RECIST v1.1)
7. WHO performance status 0 or 1
8. Age ≥ 18
9. Estimated life expectancy > 3 months.
10. Adequate bone marrow function: Haemoglobin ≥ 100 g/L, White Blood Cell ≥ 3.0 x 10^9/L, Absolute neutrophil ≥ 1.5 x 10^9/L, Platelet ≥ 100 x 10^9/L
11. Adequate liver function: Total bilirubin ≤1.5 x Upper Limit of Normal (ULN); ALT/AST and ALP≤ 2.5 x ULN or ≤ 5 x ULN if related to liver metastases
12. Adequate renal function: Serum urea and creatinine < 1.5x ULN AND Calculated creatinine clearance (GFR) ≥50 mL/min. If the calculated GFR is below 50, isotope clearance test is required to confirm GFR ≥50 mL/min
13. Electrolytes: Potassium ≥ 4.0 mmol/L and ≤ 5.5 mmol/L, Magnesium ≥ Lower Limit of Normal and ≤ 1.23 mmol/L, Corrected calcium within institution normal range
14. Negative pregnancy test for women of child-bearing potential AND be using adequate barrier contraception, which must be continued for 12 months after completion of treatment (male patients must also agree to use barrier contraception during the trial and for 12 months after completion of treatment)
15. Able to swallow oral medication
16. Capable of giving written informed consent

Exclusion Criteria:

1. Patients undergoing current treatment with curative intent
2. Previous or current malignancies of other histological types within the last 5 years (exceptions listed in the trial protocol)
3. Any prior exposure to VEGF, EGFR or RET inhibitors or history of hypersensitivity to vandetanib or any excipient agents
4. Evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
5. Evidence of active uncontrolled infection (patients on antibiotics are eligible)
6. Chronic gastrointestinal disease (e.g. Inflammatory Bowel Disease) or significant bowel resection that would preclude adequate absorption
7. Cardiovascular exclusion criteria (complete list provided in the trial protocol):

   * Significant cardiac event (myocardial infarction), New York Heart Association Class II or above, within 12 weeks before registration, or presence of cardiac disease that in the opinion of the investigator increased the risk of ventricular arrhythmia
   * Prior or current cardiomyopathy
   * Baseline LVEF < 40% as measured by ECHO/MUGA
   * Atrial fibrillation with heart rate >100 bpm
   * Unstable ischaemic heart disease (myocardial infarction within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
   * History of arrhythmia that was symptomatic or required treatment
   * QTcB prolongation >480 ms at baseline
   * QT prolongation with other medications that required discontinuation of that medication
8. Any psychiatric or other disorder likely to impact on informed consent or ability to manage isolation
9. Major surgery within 28 days prior to registration
10. Brain metastases or spinal cord compression, unless treated at least four weeks before the first dose and stable without steroid treatment for 10 days
11. Any concomitant medications that may affect QTc, induce or inhibit CYP3A4 function (with the exception of somatostatin or somatostatin analogue) and/or prohibited medications
12. Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity | From start of cycle 1 to end of cycle 1 (each cycle = 12 weeks)
  Detailed adverse event monitoring will be conducted according to CTCAE v4.03. Dose Limiting Toxicity (DLT) is defined as any adverse event or laboratory abnormality detailed in the trial protocol, that is considered to be highly probable or probable trial treatment related and commencing anytime during the DLT evaluation period (from start of cycle 1 to cycle 1 week 12). Adverse Events include: Haematological, Clinical Chemistry, Cardiovascular, Gastrointestinal, Skin.

SECONDARY OUTCOMES:
Objective response | Determined using imaging scans performed at baseline (registration), then every 3 months after start of treatment until disease progression up to 3 years from date of registration
  Response will be assessed according to RECIST v1.1. Confirmation of complete or partial response is not required. Stable disease will be considered the best response only is a second assessment has been carried out which confirmed stable disease at least 4 weeks after trial entry. Assessment will be determined using CT scans and 123I-mIBG scans performed at baseline, then every 3 months after start of treatment until disease progression (up to 3 years from registration)
Occurrence and Severity of Adverse Events | From date of registration until 30 days after completion of trial treatment (vandetanib and/or 131I-mIBG)
  Will include all grade 1-5 adverse events.
Progression Free Survival | From date of registration to date of documented disease progression or death from any cause, whichever comes first, assessed up to 3 years from date of registration
  Progression-free survival will be calculated from the date of trial entry to the date of documented disease progression, or death from any cause. Where progression is suspected and subsequently confirmed by scans, the date of documented suspected progression will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Thirlwell, Principal Investigator — University College London (UCL) Cancer Institute
Locations (3):
- United Kingdom (3):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London